CLINICAL TRIAL: NCT05568836
Title: Relationship Between Serum Vitamin D and Outcomes of Liver Transplantation in Cirrhotic Patients Undergoing Liver Transplantation and Effects of Vitamin D Supplementation in Post-transplant Period
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Prof., National Nutrition and Food Technology Institute
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 31748
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Liver Transplant; Complications; Vitamin D Deficiency
Keywords: vitamin D; liver transplantation
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): single dose of 300000 IU vitamin D injection (IM)
  Interventions: Dietary Supplement: vitamin D supplementation
- Control (Other): No intervention
  Interventions: Other: control

INTERVENTIONS:
Dietary Supplement: vitamin D supplementation — Intervention group will receive a single IM injection of 300000 IU vitamin D
  Arms: Intervention
Other: control — control group will receive nothing
  Arms: Control

SUMMARY:
The study population is patients with liver cirrhosis undergoing liver transplantation; In this study, the sample will be selected from cirrhosis patients undergoing liver transplantation in Taleghani (Tehran), Imam Khomeini (Tehran) and Abu Ali Sina hospitals(Shiraz).

This study uses the recorded information of patients with cirrhosis who have undergone liver transplantation so far and have inclusion criteria and no exclusion criteria. First, we extract demographic and clinical and pathophysiological information of patients, including age, sex, BMI, cause of cirrhosis, medical status at the time of liver transplantation, history of abdominal surgery, portal vein thrombosis, and waiting time for liver transplantation. In the next step, we examine the serum level of vitamin D in different age and sex groups and determine the prevalence of vitamin D deficiency for each group. It should be noted that in this study, the serum level of 25-hydroxy vitamin D below 20 ng/mL will be considered an insufficient level.

In the next step, in patients 12 years of age and older, according to serum bilirubin, serum creatinine, serum sodium and INR, we calculate the MELD-Na score and evaluate it with the serum level of vitamin D or 25-hydroxy vitamin D. We also use PELD scores in patients younger than 12 years of age, which consist of age, serum albumin, total bilirubin, INR, and stunted growth.

Follow-up will be done by calling the patients and recruitment every 3 month. ACR or acute cell rejection is usually suspected after elevated liver enzymes (serum aminotransferases, alkaline phosphatase, gamma glutamyl transpeptidase) or bilirubin (30). The incidence of ACR and Overall survival (OS) will be considered as the end point of the first phase of the study, and finally the incidence of 25-hydroxy vitamin D before transplantation with MELD-Na or PELD score will be examined. ACR and OS, we deal with statistical tests.

In the second phase of the study, which is a clinical trial, 50 sample patients with vitamin D deficiency will be selected from Taleghani Hospital; After transplanting, we will inject 300,000 units of vit D IM and compare their ACR and OS levels with those who have been deficient in vitamin D but whose vitamin D status has not improved. It is worth mentioning that in the second phase of the study, patients will be followed up to 3 months after liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* ESLD underwent liver transplantation
* Creatinine, bilirubin and INR measured
* Measured liver enzymes such as serum aminotransferases, alkaline phosphatase, gamma glutamyl transpeptidase / or bilirubin

Exclusion Criteria:

* People with acute liver failure
* People who have had multiple organ transplants
* Primary graft non-function (PNF) individuals

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-10 (Estimated)

PRIMARY OUTCOMES:
ACR (acute cell rejection) | at the 3rd and 6th months after transplantation
  elevated liver enzymes (serum aminotransferases, alkaline phosphatase, gamma glutamyl transpeptidase) or bilirubin

SECONDARY OUTCOMES:
MELD-Na or PELD score | at the 3rd and 6th months after transplantation
Serum vitamin D | at the 3rd and 6th months after transplantation

IPD SHARING:
Plan to Share IPD: Undecided